CLINICAL TRIAL: NCT03518372
Title: Myocardial Injury and Intraoperative Tissue Oximetry in Patients Undergoing Spine Surgery (MONITOR)
Brief Title: Myocardial Injury and Intraoperative Tissue Oximetry in Patients Undergoing Spine Surgery
Acronym: MONITOR
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: Tissue Oximetry and Troponin; IRB#14-12996 (Other: Institutional Review Board)
Record Dates: First submitted 2018-04-24; First posted 2018-05-08 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Hypoxia; Myocardial Injury; Surgery--Complications
Keywords: Hypoxia; Myocardial Injury; Surgery--Complications; Tissue Oximetry; Near-infrared Spectroscopy (NIRS)
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Biospecimen Retention: Samples With DNA — Blood samples: Plasma for high-sensitivity Troponin T analysis. Three samples in total: One baseline, one on first postoperative day and one on second postoperative day. Each samples is 4.5 mL.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myocardial injury after non-cardiac surgery (MINS) is common in patients undergoing major surgery. Many of the events are undetected and associated with a high 30-day mortality risk. Knowledge of which perioperative factors that predicts MINS is lacking. Decrease in tissue oxygenation (StO2) is common in patients undergoing major spine surgery and is associated with postoperative complications in these patients. However, an association between decrease in tissue oxygenation and MINS has not been examined. This group of patients may have other potential predictors of postoperative complications that the study group would like to investigate. In this observational cohort study, we will include 70 patients undergoing major spine surgery at University of California San Francisco. The primary hypothesis is that decrease in intraoperative tissue oxygenation is associated with postoperative myocardial injury.

DETAILED DESCRIPTION:
Significance:

Each year 10 million people worldwide suffer from myocardial injury after non-cardiac surgery (MINS). The majority of these events are undetected because they are asymptomatic and there is sparse knowledge about triggering causes. Major surgery is associated with a high risk of postoperative complications. These include covert stroke, myocardial injury and -infarction, and are all major contributors to mortality. The 30-day post-operative mortality in patients suffering from covert stroke is increased up to eight-fold compared with matched controls and is 10% in patients with MINS, which makes it a substantial public health problem. Approximately 33% of patients undergoing major spine surgery suffer from major postoperative complications, including stroke and myocardial infarction. However, knowledge is lacking regarding which perioperative factors predict myocardial injury and -infarction, covert and overt stroke, and mortality in high-risk patients such as those undergoing major spine surgery.

Measure of tissue oxygenation with near-infrared spectroscopy (NIRS) is non-invasive and uncomplicated. Tissue desaturation is common in spine surgery patients. Previous studies found that a decrease in tissue oxygenation (StO2) was associated with postoperative complications such as creatinine elevation, hypotension and prolonged hospitalization. However, current knowledge of how tissue oxygenation affects other clinical outcomes is lacking.

Thus, to address these knowledge gaps the investigators propose a cohort study to examine the association between tissue oxygenation and MINS in patients undergoing major spine surgery.

Methods This is a prospective observational cohort study. Participants are patients undergoing major spine surgery. Measurements include blood samples, non-invasive tissue oximetry and collection of general perioperative factors from the anesthesia machine. First measurements are made on the day of surgery and further measurements are conducted on the first two postoperative days. Secondary outcomes from medical records (e.g. 30-day mortality) are collected retrospectively.

Patients will be screened from Operation Room Surgery Schedule at University of California, San Francisco (UCSF) prior to surgery. The informed consent will be obtained at the preoperative area about 30-60 min prior to surgery. Eligible patients will sign a written consent form and HIPAA Authorization for study participation. If the subject is determined to have diminished or lack a capacity to consent, a surrogate/legally authorized representative will need to be present to authorize their participation in the study and complete the applicable forms as required by UCSF and Californian law.

Data from medical records are entered by certified study personnel into REDCap (a HIPAA compliant online data collection tool) to assure all data is complete and stored correctly. Included in REDCap is a data dictionary with descriptions of every individual variable. Standard Operating Procedures (SOP's) for patient recruitment and enrollment, data collection and data extraction have been created and are available. Tissue Oximetry data is collected separately with the laboratory's oximeters. After each case/study the data is uploaded to an online secure box. As all data are collected case-by-case in the course of the study, all missing data are registered immediately as missing in REDCap and will be treated as missing data in the final data analysis.

Sample size:

The sample size assessment is based on previous studies investigation tissue oximetry and clinical outcomes.

Effect size: 0.36 (SD=0.50) based on Meng et al. (Br J Anaesth. 2017 Apr 1;118(4):551-562. doi: 10.1093/bja/aex008.):

Muscle tissue oxygenation (SmO2) time weighted area under the curve (AUC) (%*min*hr-1 (SD)):

<3 complications: 1.4 (0.8) >3 complications: 1.9 (1.2) p-value: 0.07 Proportion of patients with >3 composite complications = 33% Alpha: 0.05 Beta: 0.2 (power=0.8) Sample size: 68. We expect to include 70 patients in this study.

By convention the 5% level of alpha and 20% level of beta have been used. As this study is explorative and hypothesis-testing, the investigators consider the above calculation to contain sufficient information.

Statistical analysis:

Primary analysis will be multiple regression with adjustment for age, sex and pre-existing conditions including cardiovascular disease, coronary heart disease, heart failure, diabetes mellitus and obstructive respiratory diseases. The following pre-specified potential confounders will be tested separately: age, gender, BMI, smoking status, history of coronary artery disease, congestive heart failure, stroke, transient ischemic attacks, chronic obstructive pulmonary disease, insulin therapy, hypertension, preoperative creatinine elevation above normal, and length of surgery. Since this relationship may or may not be linear, the data will first visually be assessed by plotting the estimated probability (on the logit scale) of having the outcome as a function of StO2, using a univariable logistic regression incorporating a smooth (thin-plate regression spline) term for StO2 (smoothing parameter obtained via cross-validation). The fit of each model will be assessed by the Hosmer-Lemeshow goodness-of-fit test. STATA software will be used for the statistical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years
* Patient is undergoing elective surgery of the spine
* Surgery is scheduled to last ≥ 2 hours and involve instrumentation

Exclusion Criteria:

* Patient is < 18 years
* Patient is undergoing emergent or urgent surgery
* American Society of Anesthesiologist (ASA) status > IV
* Patient is undergoing non-instrumental surgery, such as laminectomy alone
* Patient is undergoing spine surgery for tumor or infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients are undergoing spine surgery at University of California, San Francisco at the Parnassus Campus.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
High-sensitivity Troponin T elevation | Measurement done on first and second day after surgery (highest value of the two is used in the primary analysis)
  Peak value (the highest of two postoperative measurements) of high-sensitivity Troponin T (hsTnT) elevation (as assessment for myocardial injury).

SECONDARY OUTCOMES:
Myocardial injury after non-cardiac surgery (MINS) | Baseline prior to surgery (for adjustment), first and second day after surgery.
  Myocardial injury after non-cardiac surgery (MINS) assessed as a at least one postoperative hsTnT value of 14 ng/L or more. Two independent expert adjudicators will screen medical records for patients with troponin elevations for non-ischemic etiology of the elevation (e.g. sepsis or kidney failure).

OTHER OUTCOMES:
Myocardial infarction | Within 30 days after surgery
  Diagnosis of myocardial infarction from medical record
Non-fatal cardiac arrest | Within 30 days after surgery
  Diagnosis of non-fatal cardiac arrest from medical record
Transient cerebral ischemia (TCI) | Within 30 days after surgery
  Diagnosis of transient cerebral ischemia from medical record
Overt stroke | Within 30 days after surgery
  Diagnosis of overt stroke from medical record
Mortality | Within 30 days after surgery
  From medical record

CONTACTS AND LOCATIONS:
Overall Officials: Phil Bickler, MD PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Medical Center, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Meng L, Xiao J, Gudelunas K, Yu Z, Zhong Z, Hu X. Association of intraoperative cerebral and muscular tissue oxygen saturation with postoperative complications and length of hospital stay after major spine surgery: an observational study. Br J Anaesth. 2017 Apr 1;118(4):551-562. doi: 10.1093/bja/aex008. PMID 28403400
- [Derived] Bernholm KF, Meyhoff CS, Bickler P. Association between tissue oxygenation and myocardial injury in patients undergoing major spine surgery: a prospective cohort study. BMJ Open. 2021 Sep 17;11(9):e044342. doi: 10.1136/bmjopen-2020-044342. PMID 34535471